CLINICAL TRIAL: NCT02331615
Title: Feasibility of the Use of Electrical Stimulation Using tDCS to Influence Executive Abilities After Traumatic Brain Injury Patients
Brief Title: Application of Trans Cranial Direct Current Stimulation for Executive Dysfunction After Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loewenstein Hospital (Other)
Responsible Party: Principal Investigator, yaron sacher, Application of Trans Cranial Direct Current stimulation for executive dysfunction after traumatic brain injury, Loewenstein Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18-11-LOE
Record Dates: First submitted 2014-12-17; First posted 2015-01-06 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; Executive function difficulties; Transcranial direct current stimulation
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Right (Experimental): Electrode positioning will be determined according to the EEG 10-20 international system for EEG electrode placement: Right hemisphere anodal stimulation of the dorso lateral frontal area (F3), left hemisphere catodal stimulation of the dorso lateral frontal area (F4). Intensity of 1.5 mA (milliampere) for duration of 15 minutes. A total of 9 sessions: 4 sessions a week for 2 weeks.
  Interventions: Device: neuroConn_CE_DC-STIMULATOR
- left (Experimental): Electrode positioning will be determined according to the EEG 10-20 international system for EEG electrode placement: left hemisphere anodal stimulation of the dorso lateral frontal area (F3), right hemisphere catodal stimulation of the dorso lateral frontal area (F4). Intensity of mA1.5 (milliampere) for duration of 15 minutes. A total of 9 sessions: 4 sessions a week for 2 weeks.
  Interventions: Device: neuroConn_CE_DC-STIMULATOR
- sham (Sham Comparator): The stimulator will be turned on for only a very short duration of time (msec) no meaningful stimulation is believed to be administered in such a way.
  Interventions: Device: SHAM

INTERVENTIONS:
Device: neuroConn_CE_DC-STIMULATOR — right frontal anodal stimulation
  Arms: Right
Device: neuroConn_CE_DC-STIMULATOR — left frontal anodal stimulation
  Arms: left
Device: SHAM — no meaningful stimulation will be given
  Arms: sham

SUMMARY:
Traumatic brain injury (TBI) particularly affects the frontal lobes and patients often suffer from executive dysfunction and behavioral disturbances. These types of injuries often involve axonal damage to pre frontal brain areas, which mediate various cognitive and behavioral functions. Dorsolateral prefrontal circuit lesions cause executive dysfunction, orbitofrontal circuit lesions lead to personality changes characterized by disinhibition and anterior cingulate circuit lesions present with apathy. Patients who suffered traumatic frontal lobe damage often demonstrate a lasting, profound disturbance of emotional regulation and social cognition.

Weak transcranial direct current stimulation (tDCS) induces persisting excitability changes in the human motor cortex. this effect depends on the stimulation polarity and is specific to the site of stimulation. Interacting with cortical activity, by means of cortical stimulation, can positively affect the short-term cognitive performance and improve the rehabilitation potential of neurologic patients. In this respect, preliminary evidence suggests that cortical stimulation may play a role in treating aphasia, unilateral neglect, and other cognitive disorders.

Several possible mechanisms can account for the effects of tDCS and other methods on cognitive performance. They all reflect the potential of these methods to improve the subject's ability to relearn or to acquire new strategies for carrying out behavioral tasks. It was also found that Activation of prefrontal cortex by tDCS reduces appetite for risk during ambiguous decision making.

In this tDCS study the investigator uses one anode and one cathode electrode placed over the scalp to modulate a particular area of the central nervous system (CNS). The stimulation is administered via the neuroConn DC.Stimulator Serial number 0096. The DC-STIMULATOR is a micro-processor-controlled constant current source. The DC-STIMULATOR is a CE-certified medical device for conducting non-invasive transcranial direct current stimulation (tDCS) on people.Electrode positioning is determined according to the International EEG 10-20 System.

ELIGIBILITY:
Inclusion Criteria

* Ages 18-70 years.
* Traumatic Brain injured patients who were diagnosed with executive function difficulties.
* Patients who are able to cooperate and comprehend simple instructions.
* Patients who can provide informed consent after both oral and written information was given and discussed.

Exclusion Criteria:

* Pregnancy.
* Patients who sufferred a penetrating head trauma.
* Patients who underwent a frontal craniotomy
* Patients with a history of Psychiatric problems
* In cases of Severe Porencephaly at stimulation site
* Active Epilepsy or a history of seizure.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-03; Primary Completion 2017-03-21 (Actual); Study Completion 2017-03-21 (Actual)

PRIMARY OUTCOMES:
Change from baseline MindStreams-NeuroTrax MINDSTREAMS-NEUROTRAX | day 1 (twice), day 15, day 21
  Computerized tests assess brain wellness across an array of cognitive domains including: memory, executive function, visual spatial perception, verbal function, attention, information processing speed, and motor skills. The psychometric properties of the tests exploit the advantages of computerized testing, providing precise accuracy and reaction time measurements. NeuroTrax offers an unbiased, standardized, accurate and inexpensive tool with a wide range of applicability. The specific tests that will be administered are Go-No Go Response Inhibition and Visual Spatial Processing

SECONDARY OUTCOMES:
Change from baseline Behavior Rating Inventory of Executive Function- (Adult Version) BRIEF-A | day 1, day 21
  Measures an adult's views of him- or herself and captures important observer information for a comprehensive picture of the rated individual's executive functioning.
Change from baseline Wechsler Adult Intelligence Scale (WAIS-III ) | day 1 (twice), day 15, day 21
  1. The WAIS-III, a subsequent revision of the WAIS and the WAIS-R, was released in 1997. It provided scores for Verbal IQ (Intelligence quotient ), Performance IQ, and Full Scale IQ, along with four secondary indices (Verbal Comprehension, Working Memory, Perceptual Organization, and Processing Speed).

CONTACTS AND LOCATIONS:
Locations (1):
- Loewenstein Rehabilitation Center, Raanana, Israel

REFERENCES:
- [Background] Schroeter ML, Ettrich B, Schwier C, Scheid R, Guthke T, von Cramon DY. Diffuse axonal injury due to traumatic brain injury alters inhibition of imitative response tendencies. Neuropsychologia. 2007 Nov 5;45(14):3149-56. doi: 10.1016/j.neuropsychologia.2007.07.004. Epub 2007 Jul 14. PMID 17727901
- [Background] Tekin S, Cummings JL. Frontal-subcortical neuronal circuits and clinical neuropsychiatry: an update. J Psychosom Res. 2002 Aug;53(2):647-54. doi: 10.1016/s0022-3999(02)00428-2. PMID 12169339
- [Background] Cicerone KD, Tanenbaum LN. Disturbance of social cognition after traumatic orbitofrontal brain injury. Arch Clin Neuropsychol. 1997;12(2):173-88. PMID 14588429
- [Background] Fregni F, Boggio PS, Nitsche M, Bermpohl F, Antal A, Feredoes E, Marcolin MA, Rigonatti SP, Silva MT, Paulus W, Pascual-Leone A. Anodal transcranial direct current stimulation of prefrontal cortex enhances working memory. Exp Brain Res. 2005 Sep;166(1):23-30. doi: 10.1007/s00221-005-2334-6. Epub 2005 Jul 6. PMID 15999258
- [Background] Miniussi C, Cappa SF, Cohen LG, Floel A, Fregni F, Nitsche MA, Oliveri M, Pascual-Leone A, Paulus W, Priori A, Walsh V. Efficacy of repetitive transcranial magnetic stimulation/transcranial direct current stimulation in cognitive neurorehabilitation. Brain Stimul. 2008 Oct;1(4):326-36. doi: 10.1016/j.brs.2008.07.002. Epub 2008 Oct 7. PMID 20633391
- [Background] Ferrucci R, Marceglia S, Vergari M, Cogiamanian F, Mrakic-Sposta S, Mameli F, Zago S, Barbieri S, Priori A. Cerebellar transcranial direct current stimulation impairs the practice-dependent proficiency increase in working memory. J Cogn Neurosci. 2008 Sep;20(9):1687-97. doi: 10.1162/jocn.2008.20112. PMID 18345990
- [Background] Fregni F, Boggio PS, Nitsche MA, Rigonatti SP, Pascual-Leone A. Cognitive effects of repeated sessions of transcranial direct current stimulation in patients with depression. Depress Anxiety. 2006;23(8):482-4. doi: 10.1002/da.20201. No abstract available. PMID 16845648
- [Background] Fecteau S, Pascual-Leone A, Zald DH, Liguori P, Theoret H, Boggio PS, Fregni F. Activation of prefrontal cortex by transcranial direct current stimulation reduces appetite for risk during ambiguous decision making. J Neurosci. 2007 Jun 6;27(23):6212-8. doi: 10.1523/JNEUROSCI.0314-07.2007. PMID 17553993
- [Background] Beeli G, Casutt G, Baumgartner T, Jancke L. Modulating presence and impulsiveness by external stimulation of the brain. Behav Brain Funct. 2008 Aug 4;4:33. doi: 10.1186/1744-9081-4-33. PMID 18680573
- [Background] Boggio PS, Ferrucci R, Rigonatti SP, Covre P, Nitsche M, Pascual-Leone A, Fregni F. Effects of transcranial direct current stimulation on working memory in patients with Parkinson's disease. J Neurol Sci. 2006 Nov 1;249(1):31-8. doi: 10.1016/j.jns.2006.05.062. Epub 2006 Jul 14. PMID 16843494
- [Background] Jo JM, Kim YH, Ko MH, Ohn SH, Joen B, Lee KH. Enhancing the working memory of stroke patients using tDCS. Am J Phys Med Rehabil. 2009 May;88(5):404-9. doi: 10.1097/PHM.0b013e3181a0e4cb. PMID 19620953
- [Background] Monti A, Cogiamanian F, Marceglia S, Ferrucci R, Mameli F, Mrakic-Sposta S, Vergari M, Zago S, Priori A. Improved naming after transcranial direct current stimulation in aphasia. J Neurol Neurosurg Psychiatry. 2008 Apr;79(4):451-3. doi: 10.1136/jnnp.2007.135277. Epub 2007 Dec 20. PMID 18096677
- [Background] Bikson M, Datta A, Elwassif M. Establishing safety limits for transcranial direct current stimulation. Clin Neurophysiol. 2009 Jun;120(6):1033-4. doi: 10.1016/j.clinph.2009.03.018. Epub 2009 Apr 24. No abstract available. PMID 19394269
- [Background] Poreisz C, Boros K, Antal A, Paulus W. Safety aspects of transcranial direct current stimulation concerning healthy subjects and patients. Brain Res Bull. 2007 May 30;72(4-6):208-14. doi: 10.1016/j.brainresbull.2007.01.004. Epub 2007 Jan 24. PMID 17452283
- [Background] Dundas JE, Thickbroom GW, Mastaglia FL. Perception of comfort during transcranial DC stimulation: effect of NaCl solution concentration applied to sponge electrodes. Clin Neurophysiol. 2007 May;118(5):1166-70. doi: 10.1016/j.clinph.2007.01.010. Epub 2007 Feb 27. PMID 17329167
- [Background] Palm U, Keeser D, Schiller C, Fintescu Z, Nitsche M, Reisinger E, Padberg F. Skin lesions after treatment with transcranial direct current stimulation (tDCS). Brain Stimul. 2008 Oct;1(4):386-7. doi: 10.1016/j.brs.2008.04.003. Epub 2008 Jun 20. No abstract available. PMID 20633396
- [Background] Utz KS, Dimova V, Oppenlander K, Kerkhoff G. Electrified minds: transcranial direct current stimulation (tDCS) and galvanic vestibular stimulation (GVS) as methods of non-invasive brain stimulation in neuropsychology--a review of current data and future implications. Neuropsychologia. 2010 Aug;48(10):2789-810. doi: 10.1016/j.neuropsychologia.2010.06.002. Epub 2010 Jun 11. PMID 20542047
- [Background] Liebetanz D, Koch R, Mayenfels S, Konig F, Paulus W, Nitsche MA. Safety limits of cathodal transcranial direct current stimulation in rats. Clin Neurophysiol. 2009 Jun;120(6):1161-7. doi: 10.1016/j.clinph.2009.01.022. Epub 2009 Apr 28. PMID 19403329
- [Background] Iyer MB, Mattu U, Grafman J, Lomarev M, Sato S, Wassermann EM. Safety and cognitive effect of frontal DC brain polarization in healthy individuals. Neurology. 2005 Mar 8;64(5):872-5. doi: 10.1212/01.WNL.0000152986.07469.E9. PMID 15753425
- [Background] Nitsche MA, Paulus W. Excitability changes induced in the human motor cortex by weak transcranial direct current stimulation. J Physiol. 2000 Sep 15;527 Pt 3(Pt 3):633-9. doi: 10.1111/j.1469-7793.2000.t01-1-00633.x. PMID 10990547
- [Background] Nitsche MA, Niehaus L, Hoffmann KT, Hengst S, Liebetanz D, Paulus W, Meyer BU. MRI study of human brain exposed to weak direct current stimulation of the frontal cortex. Clin Neurophysiol. 2004 Oct;115(10):2419-23. doi: 10.1016/j.clinph.2004.05.001. PMID 15351385
- [Background] Nitsche MA, Paulus W. Sustained excitability elevations induced by transcranial DC motor cortex stimulation in humans. Neurology. 2001 Nov 27;57(10):1899-901. doi: 10.1212/wnl.57.10.1899. PMID 11723286
- [Background] Boggio PS, Nunes A, Rigonatti SP, Nitsche MA, Pascual-Leone A, Fregni F. Repeated sessions of noninvasive brain DC stimulation is associated with motor function improvement in stroke patients. Restor Neurol Neurosci. 2007;25(2):123-9. PMID 17726271